CLINICAL TRIAL: NCT03291613
Title: PINPOINT: Gaming Technology to Engage Adolescent Sickle Cell Patients in Precision Pain Management
Brief Title: Gaming Technology to Engage Adolescent Sickle Cell Patients in Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: HPC International, Inc. (Industry); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R43MD010746-01 (NIH); 0308 (Other: Klein Buendel, Inc.); 1R43MD010746-01 (NIH)
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Results first posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-01

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Adolescence; Pain Assessment; Tablet Application; Pain; mHealth
MeSH Terms: conditions — Anemia, Sickle Cell; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pinpoint App (Experimental): Tablet application.
  Interventions: Other: Pinpoint App

INTERVENTIONS:
Other: Pinpoint App — Tablet app with pain assessment and communication education, and pain assessment tool.

SUMMARY:
Sickle cell disease (SCD) is a common genetic disorder characterized by episodes of pain, yet assessments to identify type, intensity, frequency, and phase of pain among SCD adolescents is lacking. Research shows that interactive gaming technology can enhance adolescents' learning, and can be especially effective in delivering health-related messages and tools to improve their self-care. Pinpoint is an interactive gaming tablet app that will be developed with the significant input of clinical experts to assist SCD teens with better identification and self-report of their pain.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is the most common inherited blood disorder in the U.S. and disproportionately affects African Americans and Hispanics. Approximately, 1,000 U.S. children are born with SCD annually. SCD results from abnormal hemoglobin and causes red blood cells (RBCs) to become misshaped ("sickle-shaped"). Sickled cells can block the flow of blood in small arteries causing tissue and organ damage and other life-threatening comorbidities. SCD complications can be serious and have a significant impact upon well-being and quality of life. Pain is the hallmark symptom associated with SCD, and is the most common clinical problem seen in children and the number one cause of SCD-related hospital admissions. If left untreated, these painful episodes can result in morbidity and mortality. Accurate assessment of pain specifiers (type, frequency, and intensity of pain) can help with ameliorating pain quickly and effectively. Despite children being accurate self-reporters of their pain, strategies which are effective and engaging to assist with pain identification are lacking. Reducing barriers to collection and promoting the value of accurate SCD pain assessment is a need in pediatric medicine. Pinpoint will be an innovative interactive assessment tool that engages patients while allowing physicians to collect important health data. This project will test the feasibility of applying gamification principles to develop a tablet application ("app") for 13-17 year olds with SCD. Specifically, this Phase I SBIR project will (1) develop a Pain Assessment Tool (PAT) to describe and categorize specific types of pain experienced by adolescents with SCD; and (2) create an app ("Pinpoint"), that will translate the PAT into gamified technology. The goal of Pinpoint is to engage adolescent patients and improve pain specification by developing a game-based pain assessment tool delivered via a tablet app to engage adolescent SCD patients, improve their pain specification self-report, and improve pain management by clinicians. The PAT will be developed using expert guidance from preeminent SCD clinicians. User-centered Design theory will be applied in the development of the app and will be guided by iterative cognitive interviews and focus groups with members of the target population, SCD teens. The project specific aims are to (1) develop the PAT using guidance from an Expert Advisory Board (EAB) of SCD clinicians; (2) conduct a series of cognitive interviews with adolescent SCD patients to guide and refine PAT development; (3) conduct iterative focus groups with adolescent SCD patients to guide and refine user interface design of the Pinpoint app; (4) program a functional Pinpoint prototype; and (5) conduct usability testing of the prototype with 13-17 year old SCD patients to assess functionality, navigation, and satisfaction. This project is innovative and timely. Pinpoint will be the first tablet app to identify and translate specific pain types for SCD into a gamified app using applied gamification principles.

ELIGIBILITY:
Phone Interview, Focus Group, and Usability Inclusion Criteria:

* Be 13-17 years of age
* Be diagnosed with Sickle Cell Disease
* Able to read and speak English
* Able to assent to participate

Phone Interview, Focus Group, and Usability Exclusion Criteria:

* Not 13-17 years of age
* Not diagnosed with Sickle Cell Disease
* Unable to read and speak English
* Unable to assent to participate

Healthcare Provider Interview Inclusion Criteria:

* Be a healthcare provider to teens with sickle cell disease
* Be 18 years of age or older
* Able to read and speak English
* Able to consent to participate

Healthcare Provider Interview Exclusion Criteria:

* Not a healthcare provider to teens with sickle cell disease
* Not 18 years of age or older
* Unable to read and speak English
* Unable to consent to participate

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Myers, PhD, Principal Investigator — Klein Buendel, Inc.
Locations (2):
- United States (2):
  - Klein Buendel, Inc., Golden, Colorado
  - Hilton Publishing Company, Munster, Indiana

REFERENCES:
- [Background] Brawley OW, Cornelius LJ, Edwards LR, Gamble VN, Green BL, Inturrisi C, James AH, Laraque D, Mendez M, Montoya CJ, Pollock BH, Robinson L, Scholnik AP, Schori M. National Institutes of Health Consensus Development Conference statement: hydroxyurea treatment for sickle cell disease. Ann Intern Med. 2008 Jun 17;148(12):932-8. doi: 10.7326/0003-4819-148-12-200806170-00220. Epub 2008 May 5. No abstract available. PMID 18458271
- [Background] Cope A, Darbyshire PJ. Sickle cell disease, update on management. Paediatrics and Child Health. 2013;23(11):480-485.
- [Background] Mukerji I. About sickle cell disease.Sicklecellinfo.net Web site. Available at: http://www.sicklecellinfo.net/index.htm. Published 2004. Updated March 5, 2004. Accessed March 5, 2015.
- [Background] Bhagat VM, Baviskar SR, Mudey AB, Goyal RC. Poor health related quality of life among patients of sickle cell disease. Indian J Palliat Care. 2014 May;20(2):107-11. doi: 10.4103/0973-1075.132622. PMID 25125865
- [Background] Schnog JB, Duits AJ, Muskiet FA, ten Cate H, Rojer RA, Brandjes DP. Sickle cell disease; a general overview. Neth J Med. 2004 Nov;62(10):364-74. PMID 15683091
- [Background] Stinson J, Naser B. Pain management in children with sickle cell disease. Paediatr Drugs. 2003;5(4):229-41. doi: 10.2165/00128072-200305040-00003. PMID 12662119
- [Background] Ameringer S, Elswick RK Jr, Smith W. Fatigue in adolescents and young adults with sickle cell disease: biological and behavioral correlates and health-related quality of life. J Pediatr Oncol Nurs. 2014 Jan-Feb;31(1):6-17. doi: 10.1177/1043454213514632. Epub 2013 Dec 30. PMID 24378816
- [Background] Dampier C, Ely B, Brodecki D, O'Neal P. Characteristics of pain managed at home in children and adolescents with sickle cell disease by using diary self-reports. J Pain. 2002 Dec;3(6):461-70. doi: 10.1054/jpai.2002.128064. PMID 14622732
- [Background] Schatz J, Schlenz AM, McClellan CB, Puffer ES, Hardy S, Pfeiffer M, Roberts CW. Changes in coping, pain, and activity after cognitive-behavioral training: a randomized clinical trial for pediatric sickle cell disease using smartphones. Clin J Pain. 2015 Jun;31(6):536-47. doi: 10.1097/AJP.0000000000000183. PMID 25503599
- [Background] Dampier C, Lieff S, LeBeau P, Rhee S, McMurray M, Rogers Z, Smith-Whitley K, Wang W; Comprehensive Sickle Cell Centers (CSCC) Clinical Trial Consortium (CTC). Health-related quality of life in children with sickle cell disease: a report from the Comprehensive Sickle Cell Centers Clinical Trial Consortium. Pediatr Blood Cancer. 2010 Sep;55(3):485-94. doi: 10.1002/pbc.22497. PMID 20658620
- [Background] Crandall M, Savedra M. Multidimensional assessment using the adolescent pediatric pain tool: a case report. J Spec Pediatr Nurs. 2005 Jul-Sep;10(3):115-23. doi: 10.1111/j.1744-6155.2005.00023.x. PMID 16083431
- [Background] Franck LS, Treadwell M, Jacob E, Vichinsky E. Assessment of sickle cell pain in children and young adults using the adolescent pediatric pain tool. J Pain Symptom Manage. 2002 Feb;23(2):114-20. doi: 10.1016/s0885-3924(01)00407-9. PMID 11844631
- [Background] Lopez G, Liles DK, Knupp CL. Edmonton Symptom Assessment System for outpatient symptom monitoring of sickle cell disease. South Med J. 2014 Dec;107(12):768-72. doi: 10.14423/SMJ.0000000000000209. PMID 25502156
- [Background] Panepinto JA, O'Mahar KM, DeBaun MR, Loberiza FR, Scott JP. Health-related quality of life in children with sickle cell disease: child and parent perception. Br J Haematol. 2005 Aug;130(3):437-44. doi: 10.1111/j.1365-2141.2005.05622.x. PMID 16042695

RESULTS

PARTICIPANT FLOW:
Groups:
- Pinpoint App Usability Testing: Participants used the Pinpoint tablet app for one hour.
Period: Overall Study
Arm/Group | Pinpoint App Usability Testing
Started | 13
Completed | 12
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pinpoint App Usability Testing
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.58 (1.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 0
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: System Usability Questionnaire
Description: Ten likert-type questions assessing user-friendliness of technology. Each question has five answer options that range from "Strongly Agree" to "Strongly Disagree". Scores range from 0-100. A score of 68 or above is considered above average. All scores averaged.
Time Frame: After 1-hour usability session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pinpoint App
Number analyzed (Participants) | 12
units on a scale | 86.67 (11.56)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Pinpoint App
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/13/NCT03291613/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/13/NCT03291613/SAP_001.pdf